CLINICAL TRIAL: NCT01487499
Title: Bronchoscopic Intratumoral Chemotherapy for Small Cell Lung Cancer
Brief Title: Bronchoscopic Intratumoral Chemotherapy for Small Cell Lung Cancer (SCLC)
Acronym: SCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to enroll adequate number of participants
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLC
Record Dates: First submitted 2011-12-01; First posted 2011-12-07 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients with limited stage SCLC (Experimental): Subjects with limited stage SCLC treated sequentially with cisplatin.
  Interventions: Drug: Cisplatin
- Historical Controls (No Intervention): No intervention

INTERVENTIONS:
Drug: Cisplatin — 40 mg in 40 mL of normal saline for each of 4 bronchoscopies
  Arms: patients with limited stage SCLC

SUMMARY:
This project proposes to use bronchoscopic intratumoral chemotherapy for small cell lung cancer in two fashions:

1. to implement a prospective clinical trial to test the feasibility and efficacy of intralesional chemotherapy as consolidative therapy immediately following standard systemic chemotherapy and radiation therapy for patients with limited stage SCLC by comparing tumor growth and survival rates of the treatment group and compare the outcomes to historical controls
2. to implement a prospective clinical trial to test the feasibility and efficacy as measured by tumor growth and survival rates of intralesional chemotherapy for patients with recurrent SCLC after standard treatment.

DETAILED DESCRIPTION:
Subjects will receive standard of care treatment for SCLC with added treatment of Cisplatin injection via endobronchial ultrasound aided bronchoscopy a total of four times. Outcome measurements of tumor growth and survival will be compared to subjects receiving standard of care treatment only.

ELIGIBILITY:
Inclusion Criteria: Competent adult English speaking subjects

* With limited stage SCLC who have completed standard of care treatment who are responders with no evidence of disseminated disease other than CNS metastasis,
* With recurrent disseminated SCLC after standard of care treatment with symptoms related to central tumor obstruction,
* With recurrent limited stage SCLC with mediastinal/hilar recurrence not previously treated with intratumoral cisplatin

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria
* Subjects who, in the opinion of the investigator, are at risk undergoing a bronchoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Jantz, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Limited Stage SCLC
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Limited Stage SCLC
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Solid Tumor Growth After Completion of Interventional Bronchoscopies
Description: The Organization for Research and Treatment of Cancer Response Evaluation Criteria in Solid Tumors (RECIST) system will be used to grade the response to therapy.
Time Frame: 18 months
Population: No participants were analyzed because total enrollment numbers were too low to meet any statistical analysis.
Arm/Group | Patients With Limited Stage SCLC
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival
Time Frame: 18 months
Arm/Group | Patients With Limited Stage SCLC
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Subjects will be followed for 5 years or the remainder of the subject's life in order to determine long-term 5 year survival rates.
Time Frame: 5 years
Arm/Group | Patients With Limited Stage SCLC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Patients With Limited Stage SCLC
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No